CLINICAL TRIAL: NCT03666572
Title: Pilot of a Prebiotic and Probiotic Trial in Young Infants With Severe Acute Malnutrition
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: PR-17112
Record Dates: First submitted 2018-08-28; First posted 2018-09-12 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2019-09

CONDITIONS: Severe Acute Malnutrition
Keywords: Severe Acute Malnutrition; Young Infants under 6 months age; Microbiome; Prebiotics; Probiotics
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — lacto-N-neotetraose; Lactose

STUDY DESIGN:
Intervention Model Description: 3 treatment arms for infants with SAM
  * Placebo (Lactose)
  * B. infantis alone (Bif)
  * B. infantis + prebiotic Lacto-N-neotetraose [LNnT] (Bif+prebiotic)
  Age at enrollment
  * 2-3.9 months of age
  * 4-5.9 months of age
    1. open-label treatment arm for 18 non-malnourished primarily breastfed infants - B. infantis alone (Bif)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- B. infantis alone (Bif) in SAM infants (Active Comparator): B. infantis alone (Bif) in Severe Acute Malnourished infants
  Interventions: Other: Bifidobacterium infantis with prebiotic Lacto-N-neotetraose [LNnT]; Other: Placebo (Lactose)
- B. infantis + prebiotic Lacto-N-neotetraose [LNnT] (Active Comparator): B. infantis + prebiotic Lacto-N-neotetraose [LNnT] (Bif+prebiotic) in Severe Acute Malnourished infants
  Interventions: Other: Bifidobacterium infantis
- Placebo (Lactose) (Placebo Comparator): Placebo (Lactose) in Severe Acute Malnourished infants
  Interventions: Other: Bifidobacterium infantis; Other: Bifidobacterium infantis with prebiotic Lacto-N-neotetraose [LNnT]
- B. infantis alone (Bif) in Not SAM Infants (Active Comparator): B. infantis alone (Bif) in not Severe Acute Malnourished infants
  Interventions: Other: Bifidobacterium infantis; Other: Bifidobacterium infantis with prebiotic Lacto-N-neotetraose [LNnT]; Other: Placebo (Lactose)

INTERVENTIONS:
Other: Bifidobacterium infantis — Bifidobacterium longum subsp. infantis (EVC001)
  Arms: B. infantis + prebiotic Lacto-N-neotetraose [LNnT]; B. infantis alone (Bif) in Not SAM Infants; Placebo (Lactose)
Other: Bifidobacterium infantis with prebiotic Lacto-N-neotetraose [LNnT] — Bifidobacterium infantis with prebiotic Lacto-N-neotetraose [LNnT]
  Arms: B. infantis alone (Bif) in Not SAM Infants; B. infantis alone (Bif) in SAM infants; Placebo (Lactose)
Other: Placebo (Lactose) — Placebo (Lactose)
  Arms: B. infantis alone (Bif) in Not SAM Infants; B. infantis alone (Bif) in SAM infants

SUMMARY:
Malnutrition is an ever-present problem worldwide. It is estimated that over 18 million children under the age of 5 are affected by the most extreme form of undernutrition, severe acute malnutrition (SAM). In spite of having standardized management protocols, in many hospitals, inpatient mortality reaches up to 30%. Infectious morbidity is common among survivors. Diarrhea, severe intestinal inflammation, low concentrations of fecal short-chain fatty acids (SCFAs), and severe systemic inflammation are significantly associated with mortality in SAM. Investigators of this study have earlier shown that the gut microbiota in children with SAM is immature and is causally related to SAM.

Human milk contains between 10 and 20 g/liter of oligosaccharides (human milk oligosaccharides-HMOs) which is the third most abundant solid component after lactose and lipids. HMOs are resistant to gastrointestinal digestion in host infants, and thus the greater part of HMOs reached the colon and may act as prebiotics to shape a healthy gut ecosystem by stimulating the growth of useful microorganisms by acting as receptor analogs to inhibit the binding of various pathogens and toxins to epithelial cells. Probiotics are live organisms beneficial for a healthy life. The human digestive tract possesses a diverse microbial community throughout its extent, which supports their hosts generally for healthy living. Bifidobacterium spp. is dominant microbiota in infants who are exclusively breastfed and these infants are less likely to suffer from diarrhea. According to recent studies among the most common probiotics genera Lactobacillus and Bifidobacterium, the latter is more abundant in the gut. To carry out their functional activities, Bifidobacteria must be able to survive the gastrointestinal tract transit and persist, at least transiently, in the host. The population of Bifidobacteria in the gut community drastically decreases after weaning. Certain Bifidobacteria possess the metabolic capabilities to break down the HMOs. Consequently, it is observed that HMOs support the growth of select Bifidobacteria in the gut of the infant.

Research done at icddr,b and Washington University indicates that gut microbes are related to undernutrition and that children with SAM have gut dysbiosis that mediates some of the pathologies of their condition. The standard of care in these children should be reinforced by an intervention that corrects the gut dysbiosis, improves weight gain during nutritional rehabilitation, and reduces infectious morbidity. Investigators do not have any published data on the microbiome response to probiotic supplementation (with and without prebiotics) in malnourished infants or preserving the microbiome with probiotics in non-malnourished children.

A short-term pilot study should be conducted to evaluate the microbiome response to probiotic supplementation (with and without prebiotics) in malnourished populations to justify a larger study of clinical outcomes. Additionally, non-malnourished infants who are hospitalized for infectious conditions face challenges related to gut dysbiosis caused by antibiotic usage. Here the investigators will evaluate the ability of a probiotic intervention to rescue the microbiome of primarily breastfed non-malnourished infants.

Intervention: Bifidobacterium longum subspecies infantis (EVC001) with and without prebiotic supplementation for 28 days.

Objectives: To evaluate the microbiome response to probiotic supplementation (with and without prebiotics) in infants under 6 months with severe acute malnutrition and to compare the microbiome response with healthy infants with a probiotic.

Methods: Single-blind RCT, stratified randomization will be based on infant age at the time of transfer to the Nutritional Rehabilitation Unit (NRU).

3 treatment arms for infants with SAM

1. Placebo (Lactose)
2. Bifidobacterium infantis alone (Bif)
3. Bifidobacterium infantis + prebiotic Lacto-N-neotetraose [LNnT] (Bif+prebiotic) Age at enrollment

   1. 2-3.9 months of age
   2. 4-5.9 months of age 1 open-label treatment arm for 18 non-malnourished primarily breastfed infants: Bifidobacterium infantis alone (Bif)

Population:

1. Group 1 (SAM): Infants between 2 and <6 months old with SAM as defined by weight-for-length Z score < -3 either sex, caregiver willing to provide consent for enrolment of the infant, caregiver willing to stay in the NRU for about 15 days, residence within 15 km from icddr,b
2. Group 2 (non-malnourished): Non-malnourished infants (WLZ ≥ -1) <6 months old who are hospitalized for treatment with antibiotics for the infection, infants receiving at least 50% of nutritional intake from breast milk at the time of hospitalization, either sex, residence within 15 km from icddr,b

Primary Outcome measures/variables:

Bifidobacterium infantis colonization measured by qPCR during and after supplementation (with and without prebiotics)

DETAILED DESCRIPTION:
Specific Objectives:

To evaluate the microbiome response to probiotic supplementation (with and without prebiotics) in under 6 months infants with severe acute malnutrition and to compare the microbiome response with healthy infants supplemented with probiotic.

Study Site: The study will be conducted at Dhaka Hospital of the International Centre for Diarrheal Disease Research, Bangladesh (icddr,b). The institution possesses well equipped clinical care as well as laboratory facilities capable of performing all the clinical tests.

Study population:

Group 1 (SAM) Group 2 (non-malnourished)

Intervention:

Bifidobacterium longum subsp. infantis (EVC001) with and without prebiotic supplementation for 28 days will be provided in the study.

There are several studies in the developing world where prebiotic and probiotic were used in severe acute malnutrition and among at risk infants. Safety of Bifidobacterium longum subsp. infantis (EVC001) is evident from published literature as well as safety reports (Smilowitz et al., 2017; Sheridan et al., 2017; Grenov et al., 2017; Panigrahi er al., 2017; Kerac et al., 2009). The IMPRINT Study, a Phase I clinical trial, determined the safety and tolerability of supplementing breastfed infants with B. infantis (EVC001) (Smilowitz et al., 2017). Safety of prebiotic (LNnT) was evaluated by EFSA (European Food Safety Authority) Panel on Dietetic Products, Nutrition and Allergies (NDA) related food and panel concluded that LNnT is safe for infants. The International Scientific Association for Probiotics and Prebiotics (ISAPP) recommended that an attractive target for clinical interventions will lead to new approaches that combat malnutrition (Sheridan et al., 2017). A study held in Uganda using probiotic In hospitalized SAM children revealed that probiotic may have a role in follow up of hospitalized children with SAM in outpatient phase as it showed significant reduction of diarrheal duration (Grenov et al., 2017). In rural India significant reduction was observed for culture-positive and culture-negative sepsis and lower respiratory tract infections in infants with use of symbiotic (Kerac et al., 2009). The PRONUT study did not demonstrate any case of probiotic related bacteraemia . The response of microbiota to probiotics may differ by diet or geography.

Trial arms:

3 treatment arms for infants with SAM:

* Placebo (Lactose)
* B. infantis alone (Bif)
* B. infantis + prebiotic Lacto-N-neotetraose [LNnT] (Bif+prebiotic) Each arm will be assigned to receive the standard of care diet (F-75 during the acute phase treatment of SAM, F-100 during hospital stay for nutritional rehabilitation, and standardized infant formula upon discharge). Randomization for treatment allocation will be done in 1:1 ratio using stratification by age (2-3.9 months vs. 4-6 months) to ensure equal participation of infants by age groups. Allocation will be achieved by using random permuted blocks size of 3. In total 54 participants will be enrolled with 18 infants (9+9) allocated in each treatment arm.

Prebiotic will be used in the form of LNnT (Lacto-N-neotetraose, which is produced by fermentation and is chemically identical to LNnT present in human breast milk. LNnT contains a specific linkage that B. infantis can break down while other bacteria cannot. In the in vitro assay, when the growth media contains 50% or more of LNnT, growth of B. infantis is supported, but growth of Bacteroides and E.coli is inhibited. The distribution of the glycosylhydrolases needed to consume this structure are rare among Proteobacteria (including Campylobacter) as a whole, and absent among Bacteroides and therefore LNnT should not contribute to cross feeding, even in the absence of B. infantis engraftment.

The aim of selecting the non-malnourished children is to see whether the disrupted microbiota of SAM infants recovers to higher level of B. infantis, similar to those levels seen in healthy breast fed infants who have an acute illness and are treated with an antibiotic.

Sample size:

For the pilot, we will have 18 infants per treatment arm, a total of 54 SAM infants. We will also enroll 18 non-malnourished infants for the open-label B. infantis treatment. A total of 72 infants will be the study population for this pilot.

Even if study participants drop or develop any hospital acquired infection or deteriorate, we have to complete 18 evaluable cases in each arm.

Baseline data collection procedure: All SAM and non-SAM children within the defined age groups will be screened for study eligibility criteria by the study physician. Parents / attending care givers of those fulfilling the eligibility, in application of the inclusion and the exclusion criteria, will be invited to provide their consent for enrollment of their children in the study. Upon signing a written informed consent, after providing information about the study and its interventions, explaining possible benefits and risks, and voluntary nature of participation along with the right to withdraw children at any time after the initial consent without providing any reason, children will be enrolled by the study physician. Clinical Record Form will be used to collect relevant information such as medical history including nature and duration of illness, medication for current illness; socio-demographic characteristics such as age, sex, religion, parental age with education, parents occupation, fuel use and smoking history, monthly family income, number of siblings,etc. Information would also be collected about child's feeding practice such as history of breast feeding, formula or other complementary feeding, and immunisation status; family history of tuberculosis, recent respiratory tract infection of any family members and past medical history of child would be recorded.

For long term follow up separate CRF will be used to collect information on weight, height, MUAC, feeding and co-morbidity history. Field Research Assistants will visit the houses of enrollees and will collect required information after taking written consent from parents or caregiver.

Management:

Group 1 (children with SAM): Eligible SAM infants will be treated for the stabilization phase in the Longer Stay Unit of the Dhaka Hospital of icddr,b. The standardized treatment protocol for children with SAM and diarrhea (developed at icddr,b and aligned to the WHO guidelines; Ahmed et al Lancet 1999) will be followed. Key elements include initially 2 hourly feeding with F-75 (the recommended starter formula, 130 ml/kg per day), folic acid, vitamin A, Ampicillin plus Gentamicin, temperature and blood glucose monitoring and control. Prior to initiation of antibiotics, baseline stool samples will be obtained (by fecal catheter if needed).

The stabilization phase lasts on an average 4 days in our experience. Completion of stabilization phase is characterized by a satisfactory appetite, no need for nasogastric tube feeding, good general clinical condition, absence of diarrhea, dehydration, fever, hypothermia or tachypnea.

Infants who are stabilized are transferred to the NRU upon receiving written consent from the caregiver. Stabilized infants will be randomized to the 3 treatment arms once they have completed the 5-7 day course of antibiotics. The Senior Dietician of the Hospital prepares the diet (F-100) and supplies to the NRU. F-100 is dispensed at 130 ml/kg per day every 2 hours for the first 2 days, and thereafter given every 3 hours and gradually increased by 10 ml at each serving until some feed is left. Breast feeding is encouraged in between the feeds. Amount of breast milk consumed will be estimated by test weighing of infants.

Caregivers will be trained to provide psychosocial stimulation to the infants, an activity that is done routinely in the NRU. This is done through talking or singing to the infants, age specific physical activity and play with local toys.

Measurement of breast milk intake by test weighing folloing standard published method (Islam et al., 2006):

Collection of breast milk:

Since this study will investigate the engraftment of Bifidobacteria which is linked with availability of HMOs in breast milk, we will collect 10 ml of breast milk under aseptic condition and will be analyzed for HMO content.

This analysis will be performed in laboratories that have a track record of performing these assays.

Additionally, we will also perform microbiota analysis of collected breast milk samples. This is because breast milk microbiota is likely to influence the colonization by other organisms and the intestinal mileage of infant.

Breast milk will be collected from the breast between 0700 and 1100 hr, and women will be asked to have not to fed or expressed from the study breast for at least 2 hours prior to sample collection. Before sample collection, the breast will be cleaned with an iodine swab. A complete breast expression will be collected using a single-use, sterile, collection kit (Hygienikit®; Ameda, Cary, IL, USA) and an electric breast pump (Model SMR-B-R; Ameda-Egnell, Inc.). Milk will be immediately placed on ice.

Bif (8 billion CFU/daily single dose-), Bif (8 billion CFU/daily single dose-) + Prebiotic (1gm/6hourly-4gm/day), and placebo (lactose 625mg) will be available in powder format in sachets contained within feeding kits marked with unique code numbers that match the randomization code of each infant. The sachet contents will be administered to an infant once every day for Bif and placebo sachets mixed with 5ml infant formula or breast milk and each preparation of 200ml F-100 one prebiotic (LNnT) sachet will be dissolved. Caregivers, but not study staff, will be blinded to treatment assignment.

The dose and dispensing of LNnT will ultimately be derived upon the review of recent literature as well as experience of experts working in this field. The goal is to stimulate as much as possible the natural conditions of availability of HMOs in breast milk.

The feeding kits (sachets) that have been assigned to randomized infants will be refrigerated or stored frozen until used while the participant is hospitalized. Feeding kits that have not yet been assigned to an infant will be stored in a hospital freezer with continuous temperature monitoring. The probiotic stored in the freezer (-20°C ± 5°C) can be used up until the expiration date printed on the sachet (1 year from date of packaging). It can be stored up to 31 days in the refrigerator (4°C ± 5°C). The prebiotic (LNnT) is stable at room temperature, but can be stored in the refrigerator or freezer with the probiotic.

Group 2 (non-malnourished children): Eligible non-malnourished infants will be treated as per hospital protocol. In brief, they are admitted to the Longer Stay Unit or if necessary to the ICU. The hospital has defined treatment protocols for acute watery diarrhea, pneumonia and severe pneumonia, persistent diarrhea, severe sepsis, electrolyte disorders, and hospital-acquired infections. Children will be treated at the hospital per these protocols. Exclusively breastfed infants will continue on breast milk. Others are supplemented with modified infant formula every 2-3 hours. Amount of breast milk consumed will be estimated by test weighing of infants. Treatment with Bif will start on the day of completion of the antibiotic course and will be provided to infants in the same manner as Group 1. The sachet contents will be mixed with a teaspoon of infant formula or breast milk and fed to the infant.

Even if study participants drop or develop any hospital acquired infection or deteriorate, we have to complete 18 evaluable cases in each arm.

Discharge from Hospital:

The discharge will be done if the infant with SAM has achieved a weight-for-length >-3, if possible ≥ -2 Z-score, and in case of edematous malnutrition when edema resolves and when the infant thriving and clinically well. Non-malnourished infants will be discharged when they fulfill the hospital discharge criteria.By then the caregivers will have been trained for food and supplement preparation and administration.

Follow up:

Infants with SAM will be followed up through home visits by Research Assistants twice every week until 8 weeks post randomization. Non-malnourished infants will be followed through home visits twice every week until the supplementation is complete and then once every week until 6 weeks post randomization. During such visits, the rations of infant formula (for SAM infants) and supplements (both groups) will be replenished, actual intake of the diet will be observed or the amount given and the method of reconstitution verified, and morbidity recorded on a customized case record form. Because the B. infantis supplement should be kept cool to maintain optimum viability, Research Assistants will bring the supplement to home visits in insulated boxes or coolers with ice or frozen gel packs. Although the supplement will likely warm to room temperature between visits, it is not expected that the viability loss will significantly impact the colonization of B. infantis in the gut. A miniature fridge will be provided to each participant for the study period and each parent will be instructed to keep the supplement in these containers until use.

Infants who have not yet achieved a weight-for-length ≥ -1 Z-score by 8 weeks post randomization (end of home visits) may continue to bring the infant to icddr,b for weighing and measuring and to pick up the formula rations on a routine basis until a weight-for-length ≥ -1 Z is achieved.

A long term follow up will be carried out to assess the anthropometry of enrolled participants.

Sample collection:

Fecal samples will be collected as follows.

* Stool swabs (for microbiome analysis) (13times in SAM, 11 times in non-SAM)

  * At admission, prior to antibiotic treatment
  * After stabilization, prior to randomization and supplementation
  * Day 2 of supplementation
  * Day 4 of supplementation
  * Day 7 of supplementation
  * Day 10 of supplementation (or last day in NRU if discharged sooner)
  * Day 14 of supplementation (in NRU or picked up by research assistant at home visit)
  * Day 21 of supplementation (picked up by research assistant at home visit)
  * Day 28 of supplementation (picked up by research assistant at home visit)
  * 1 week post supplementation (picked up by research assistant at home visit)
  * 2 weeks post supplementation (picked up by research assistant at home visit)
  * 3 weeks post supplementation (picked up by research assistant at home visit): SAM only
  * 4 weeks post supplementation (picked up by research assistant at home visit): SAM only
* Stool chunks or catheter fecal samples (for pH and inflammatory markers) in hospital [SAM infants only]:

  * At admission, prior to antibiotic treatment
  * After stabilization, prior to randomization and supplementation
  * Day 7 of supplementation'
  * Day 10 of supplementation (or last day in NRU if discharged sooner)
  * Day 28 of supplementation (collected by research assistant at home visit)
  * 4 weeks post supplementation (collected by research assistant at home visit)
* Stool chunks or catheter fecal samples (for pH and inflammatory markers) in hospital [non-malnourished infants only]:

  * At admission, prior to antibiotic treatment
  * After start of supplementation, at hospital discharge
  * Day 28 of supplementation (collected by research assistant at home visit)
  * 2 weeks post supplementation (collected by research assistant at home visit)

Stool sample collection in the hospital:

All children will be screened from Dhaka Hospital, icddr,b according to the above mentioned inclusion and exclusion criteria. Research staff will screen these children before administration of an antibiotic. Before collection of stool samples written consent will be taken from legal guardian.

Stool should be freshly collected from each child. The samples must be immediately aliquoted into pre-labelled 2 ml cryovials and into the shipper (~-70⁰C) as quickly as possible after collection, ideally less than 15 minutes after collection. After collection and prior to aliquoting, the stool collection vessel should be maintained on (wet) ice. Ideally the cryovials would be filled to approximately 2/3 full. Two times in a week these cryopreserved samples will be transported to Biosafety Level Laboratory in icddr,b Dhaka Hospital for storage in -80⁰C freezer. In order to prevent thawing, vials will be transferred from the shipper to the -80⁰ freezer as quick as possible while transferring to freezer boxes. These freezer boxes will not be removed from the -80⁰ freezer until they are handed over to World Courier for shipment to USA.

Measures to ensure best possible recovery of bacteria and their viability:

1. The shippers should be fully charged before the collection day and a record will be maintained for the number of times they will be opened.
2. The shippers need around 12 hours after adding liquid nitrogen to become fully charged. Therefore, we will re-charge (fill) the shippers at the end of each day and then pour off any remaining unabsorbed liquid nitrogen the next morning before using them.
3. Shippers will be weighed before charging, after charging (ie. the next morning after pouring off any unabsorbed N2), and then again at the end of each day, to know how much liquid nitrogen remains in the canister. This will allow us to estimate how much liquid N2 is needed every time we recharge and how frequently this is needed.

Stool swab collection in the Hospital and from the Community:

Stool samples will be collected as mentioned in the time schedule. Once participants are discharged from the NRU, the stool swab will be collected within a two day window of the scheduled time.

For collection of stool, child's/participant's primary caretaker will be informed one day before planned stool collection. A trained research staff will collect the first available fresh stool sample from the child on the day of the scheduled sampling.

During collection in the Hospital and in the community, the research staff will be provided with the labeled stool swab tubes (containing stabilization buffer), individually wrapped swabs (with breakpoint), a cryogenic marker, and plastic bags.

In the Hospital, the mothers/caretakers will be instructed to notify the research staff as soon as the child defecates. Then the research staff will do the following:

* Swab the baby's soiled diaper, collecting enough stool sample to entirely coat the head of the swab.
* Place the swab into the appropriately labeled green-topped collection tube and snap the swab head off at the breakpoint - the swab head will remain in the tube.
* Seal the tube tightly and shake vigorously to ensure distribution of the stool within the stabilization buffer.
* Using the provided cryogenic marker (https://www.thermofisher.com/order/catalog/product/4000221), write the date the stool was collected on the label on the tube.
* Repeat the swabbing with a second clean swab and the duplicate green-topped tube.
* Place green-topped tubes back in the provided plastic bags and store at room temperature until picked up by the health worker.

Information about antibiotic intake will be collected for each participant during the study. At the time of each sample collection, we will ask mother or other caregiver for any illness during last 14 days, and whether treated. The nature of medicine will be verified by physical inspection of the medicine, the prescription and by asking the name or if the medicine was a powder that had to be reconstituted.

Saliva sample collection from mother:

We will do the "Secretor status phenotyping assay" in mothers' saliva to see the secretor status of mothers to detect HMO status as well as link with the Microbiota of infants.

Saliva sample collection procedure

1. Mothers' should wash the hands and rinse the mouth with cold water, and spit water out completely.
2. They will remove the sampler being careful to touch only the handle.
3. Mother will hold the handle Oracle sampling tube as a toothbrush and will insert in her mouth and will rub a sponge against her gums for one minute. Ensure that the sponge is completely saturated.
4. without touching the sponge, they will insert the sampler into the original Oracol tube, sponge down, and will close the lid tightly.
5. Mother will give the Oracle sampler tube back to the study staff (who will label and refrigerate the tubes if the samples will not be processed on the same day).

Collection and transport of fecal samples from the community Each trained community health worker will be responsible for certain number of stool collections per month. She will contact mother over cell phone and arrive at the child's house early in the morning with a bench top nitrogen shipper and collect the stool swab.

Initial collection of fecal samples should be made in a suitable sterile container after which smaller aliquots of fecal material should be transferred by the field worker (within 20 minutes of defecation) into pre-labeled, sterile 2ml cryo-safe tubes. Tube labels should minimally include the Participant's Sample ID (SID) and the date of collection.

Wearing clean, disposable latex gloves, the health workers will fill each 2 ml cryo-vial approximately one-half to two-thirds full using a sterile spatula and cap tightly. Any buffers, preservatives or additives will not be added to the sample. Precaution will be taken during use of screw cap vials and not overfilling them as this will minimize the potential for cross-contamination of samples during transport and storage.

Then they will place the capped vials into liquid nitrogen pre-charged 'dry shippers' immediately to transport back to the laboratory. Although difficult, the specimens should be transferred to dry shippers within 20 minutes of defecation. In the laboratory, trained staff will empty the vials from the dry shipper into a bucket of dry ice to prevent thawing while sorting and transferring the vials to 9x9 freezer boxes for longer term storage and transport.

Reporting:

Information will be recorded on Stool Field Collection Form (SFC).

Investigations:

Tests performed at icddrb:

* determining fecal pH in hospital lab
* Testing of Myeloperoxidase and other biomarker levels in fecal samples

Tests performed by Evolve Biosystems:

* Next Generation Sequencing, Metagenomics and q PCR analyses of samples
* Immune- related tests- Multiplex analysis of inflammatory and immune-related cytokines/analytes
* IL-10, TGF beta, IL-2, TNF alpha, IL-17, IL-22, IL-8, IL-6, IP-10
* ELISAs for sCD83, sTLR2 and fecal lipocalin 2

Stool PH:

Stool PH will be measured to assess the change from baseline in stool pH during supplementation.

Myeloperoxidase:

Myeloperoxidase is a specific marker of neutrophil activity. It was chosen because it is not elevated in breast milk or in the stools of breastfed children as are lactoferrin and calprotectin (Dorosko et al., 2008) and stool MPO levels have been correlated with disease activity in inflammatory bowel disease as assessed both by endoscopic and biochemical parameters (SAIKI T, 1998). MAL-ED study has already demonstrated the role of MPO as a marker of gut function (McCormick et al., 2017).

We will measure this biomarker concentration by a commercial ELISA.

Next Generation Sequencing: In recent years, several next-generation sequencing technologies have been established (Shendure & Ji, 2008) which further make it possible to analyze a large number of microorganisms in different environments (Tringe et al., 2005) and human body sites (Ding & Schloss, 2014, including the human gut (Methé et al., 2012).

16S rDNA sequence analysis and metagenomics are two effective DNA sequencing techniques, and both have been used to study uncultivated gut microbial communities. 16S rDNA sequence analysis focuses on the sequencing of the conserved 16S rDNA gene present in all microbes (Woese & Fox, 1977) and has established a series of novel connections between intestinal microbiota composition and disease (Blaser et al., 2013). The research based on 16S rDNA sequence is a technique to reveal "who's there?" in a given microbial community, while shotgun metagenomic sequencing will be able to answer the complementary question of "what can they do?" (Lepage et al., 2012). Next generation sequencing will be performed to detect the engraftment of organism especially B. infantis after intervention in severely malnourished infants and comparing it with well nourished children.

Metagenomics:

Metagenomics was first described in 1998 by Handelsman and Rodon ( Handelsman et al., 1998) and became another DNA sequencing approach to study the complex gut microbial community. It aims to catalog all the genes from a community by the random sequencing of all DNA extracted from the sample (Qin et al., 2010). Firstly, the total DNA of all microorganisms is extracted from fecal samples. Before being sequenced, total DNA samples are randomly sheared by a "shotgun" approach. The comprehensive sequences are then analyzed to obtain either species profiles based on phylogenetic markers (16S rDNA) (Sunagawa et al., 2010) or genomic profiles based on whole genomes (Tringe et al., 2005). Metagenomics plays a role in understanding the human gut microbiome, including the diversity of the gut microbiome, identifying novel genes, and determining the etiology of functional dysbiosis (Wang et al., 2015). Baseline composition of gut microbiota (metagenomic analysis) and Bifidobacterium colonization (relative abundance) by metagenomic analysis during/after supplementation will be done.

qPCR: Real time PCR will be done for quantitative detection of organism in DNA directly extracted from stool sample. B. infantis colonization by qPCR during and after supplementation (with and without prebiotics) will be done.

Cytokines:

Any cytokine that is produced locally as a result of gut inflammation may leak into the bowel lumen and appear in the stools. Large inflammatory infiltrate in the diseased mucosa of gut causes raised cytokines in stool. We will do cytokine assays to detect gut inflammation. We will measure in stool samples Interleukin-10 (IL-10), Transforming Growth Factor-β (TGF-β), Interleukin-2 (IL-2), Tumor Necrosis Factor-α (TNF-α), Interleukin-17 (IL-17), Interleukin-22 (IL-22), Interleukin-8 (IL-8), Interleukin-6 (IL-6), Interferon Gamma-Induced Protein 10 (IP-10).

ELISAs for sCD83, sTLR2:

A soluble form of CD83 is released from activated dendritic cells and B lymphocytes, and is detectable in normal human sera (Hock et al., 2001). Toll-like receptors (TLRs) are a class of pattern recognition receptors (PRRs) that play a key role in innate immunity and trigger a specific immune response. sTLR2 has been detected in human fluids, such as plasma, breast milk, saliva and amniotic fluid as well as in supernatant of cultured monocytes (LeBouder et al., 2003; Kuroishi et al., 2007; Dulay et al., 2009) We will isolate sCD83 and sTLR2 from stool samples of malnourished infants.

Fecal lipocalin 2:

This glycoprotein is expressed in several cells and, has been associated with primary and secondary granules of human neutrophils (Roudkenar et al., 2007). Upregulation of Lcn-2 is observed in tissue damaging conditions such as infection, kidney injury, cancer, ulcerative colitis and burn injury where production of free radicals occurs (Chassaing et al., 2012). Lipocalin-2 correlates less tightly with the neutrophil markers, it may provide a complementary marker of epithelial cell disruption or damage ( Prata et al., 2016). We will do the test for both the malnourished and well nourished infants to detect enterocyte damage.

Breast milk microbiota and HMO analysis:

There are several study where breast milk analysis (Williams et al., 2017) and bacterial community in breast milk (Hunt et al., 2011) were assessed. In this study Microbiota analysis will be done with 16S rDNA sequence analysis. HMO measurement will be done to know LnNT level.

Data processing Procedure:

* Questionnaires will be visually scanned soon after interview & marked for omissions, inconsistencies or mistakes that will be addressed immediately
* SPSS will be used & data will be entered after creating a template for each data entry file with appropriate logical and consistency checks
* Data will be continuously entered as the data are being generated in hospital and laboratory
* Data will be validated by a series of logical and range checks, producing summary statistics and tables
* In addition 50 % CRF (and all variables) will be checked by investigator(s).
* Data will be immediately copied on the hard disks of two computers as soon as data verification will be completed.

Sample Size Calculation and Outcome (Primary and Secondary) Variable(s):

For the pilot study, we will enrol 18 SAM infants per treatment arm, and additional 18 non-malnourished children, thus a total of 72 infants.

Data Analysis Data will be entered in to the pre-tested Clinical Record Forms (CRFs) using SPSS (20.0 version, Armonk, NY) and finally cleaned with repeated check. To know the outcome of prebiotic and probiotic supplementation in our study children for normally distributed data we will perform ANOVA and in case of non-normal distribution of measurements, equivalent non-parametric tests like Kruskal-Wallis H test will be used and appropriate post hoc test will be done for the sub-group analysis, if required. A probability of less than 0.05 will be considered as statistically significant and strength of association will be determined by calculating odds ratio (OR) and 95% confidence intervals (CI). If any death occurs we will perform verbal autopsy and evaluate the associated factors of death by the same analytic plan.

Data Safety Monitoring Plan (DSMP) Data safety Monitoring will be rigorously performed throughout the course of the study. All forms will be reviewed by study physician after enrolment and data collection followed by supervisor for completeness, legibility, and internal consistency. Administration of prebiotic and probiotic in hospital will be in presence of study physician. All aspects of specimen accession, processing and interpretation will also be performed according to SOPs.

Collaborative Arrangements icddr,b will perform the study in collaboration with Evolve BioSystems, Inc. USA , a private enterprise established in California by internationally reputed academicians researching into infant gut microbiome and its critical association with human breast milk.

ELIGIBILITY:
Inclusion Criteria:

Group 1 (SAM):

* Infants between 2 and <6 months old with SAM as defined by weight-for-length < -3 Z and/ or bilateral pedal edema
* either sex
* caregiver willing to provide consent for enrolment of the infant
* caregiver willing to stay in the Nutritional Rehabilitation Unit for about 15 days
* residence within 15 km from icddr,b

Group 2 (non-malnourished):

* Non-malnourished infants (WLZ ≥ -1) <6 months old who are hospitalized for treatment with antibiotics for infection (infants who come with a history of antibiotic intake for 3 days or more will be eligible; the last dose of such an antibiotic will have to be taken within last 24hours, the antibiotic intake should be documented by the verification of a prescription, the bottle of antibiotic or asking the caregiver about the name of antibiotic or its price and how it is reconstituted)
* infant receiving at least 50% of nutritional intake from breast milk at the time of hospitalization
* either sex
* residence within 15 km from icddr,b

Exclusion Criteria:

* Septic shock or very severe pneumonia requiring assisted ventilation
* acute kidney injury on admission
* congenital defects interfering with feeding such as cleft palate
* chromosomal anomalies
* jaundice
* tuberculosis
* presence of bilateral pedal edema ongoing maternal antibiotic usage for breastfeeding infants

Group 1 (SAM) additional exclusion criteria:

Infants receiving ≥75% of nutrition from breast milk

Group 2 (non-malnourished) additional exclusion criteria:

Infants receiving <50% of nutrition from breast milk

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2018-09-21 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Number of colonization of Bifidobacterium infantis in the intestine of the study participants as measured by qPCR during and after 28 days of supplementation (with and without prebiotics) | 28 days
  Number of colonization of Bifidobacterium infantis in the intestine of the study participants as measured by qPCR during and after 28 days of supplementation (with and without prebiotics)

SECONDARY OUTCOMES:
Baseline composition of gut microbiota of the study participants as estimated by metagenomic analysis | 28 days
  Baseline composition of gut microbiota of the study participants as estimated by metagenomic analysis
Bifidobacterium colonization (relative abundance) estimated by metagenomic analysis during/after supplementation of 28 days | 28 days
  Bifidobacterium colonization (relative abundance) estimated by metagenomic analysis during/after supplementation of 28 days
Colonization of naturally occurring Bifidobacterium infantis strains identified by qPCR | 28 days
  Colonization of naturally occurring Bifidobacterium infantis strains identified by qPCR
Baseline stool pH | At screening
  Baseline stool pH
Change from baseline in stool pH during supplementation for 28 days | 28 days
  Change from baseline in stool pH during supplementation for 28 days
Composition of breast milk microbiota | 28 days
  Composition of breast milk microbiota
Breast milk Human Milk oligosaccharide contents | 28 days
  Breast milk Human Milk oligosaccharide contents
Rate of body weight gain (g/kg per day) by the study participants (Secondary clinical outcome for Severe Acute Malnourished infants) | 8 weeks
  Rate of body weight gain (g/kg per day) by the study participants
Morbidity during Nutrition Rehabilitation Unit stay and post-discharge including number of (Secondary clinical outcome for Severe Acute Malnourished infants) | 8 weeks
  Morbidity during Nutrition Rehabilitation Unit stay and post-discharge including number of episodes requiring re-hospitalization
Recovery from Severe Acute Malnourished state by the infants as measured by absence (Secondary clinical outcome for Severe Acute Malnourished infants) | 2 weeks (approximated)
  Recovery from Severe Acute Malnourished state by the infants as measured by absence of bi-pedal edema and or achievement of Weight-for-Length Z-score ≥ -2
Recovery from moderate acute malnutrition (MAM) measured by achievement of Weight-for-Length Z-score ≥ -1 (Secondary clinical outcome for Severe Acute Malnourished infants) | 8 weeks
  Recovery from moderate acute malnutrition (MAM) measured by achievement of Weight-for-Length Z-score ≥ -1
Length-for-age Z score measured by length (Secondary clinical outcome for Severe Acute Malnourished infants) | 8 weeks
  Length-for-age Z score measured by length
Fecal Myeloperoxidase levels (Secondary clinical outcome for Severe Acute Malnourished infants) | 28 days
  Fecal Myeloperoxidase levels.
Duration of hospital stay (Secondary clinical outcome for Not Severe Acute Malnourished infants) | Through study completion, an average of 2 weeks
  Duration of hospital stay
Re-hospitalization rates (Secondary clinical outcome for Not Severe Acute Malnourished infants) | 6 weeks
  Re-hospitalization rates
Fecal Myeloperoxidase levels. (Secondary clinical outcome for Not Severe Acute Malnourished infants) | 28 days
  Fecal Myeloperoxidase levels.
Etiology of diarrhea in young infants by TAC assay | 28 days
  Etiology of diarrhea in young infants in this study by TAC assay
Change of anthropometry in long term follow up | 20 months
  Anthropometry will be collected from study completed participants

CONTACTS AND LOCATIONS:
Overall Officials: Tahmeed Ahmed, MBBS, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Dhaka Hospital, International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chassaing B, Srinivasan G, Delgado MA, Young AN, Gewirtz AT, Vijay-Kumar M. Fecal lipocalin 2, a sensitive and broadly dynamic non-invasive biomarker for intestinal inflammation. PLoS One. 2012;7(9):e44328. doi: 10.1371/journal.pone.0044328. Epub 2012 Sep 5. PMID 22957064
- [Background] Ding T, Schloss PD. Dynamics and associations of microbial community types across the human body. Nature. 2014 May 15;509(7500):357-60. doi: 10.1038/nature13178. Epub 2014 Apr 16. PMID 24739969
- [Background] Dulay AT, Buhimschi CS, Zhao G, Oliver EA, Mbele A, Jing S, Buhimschi IA. Soluble TLR2 is present in human amniotic fluid and modulates the intraamniotic inflammatory response to infection. J Immunol. 2009 Jun 1;182(11):7244-53. doi: 10.4049/jimmunol.0803517. PMID 19454721
- [Background] Grenov B, Namusoke H, Lanyero B, Nabukeera-Barungi N, Ritz C, Molgaard C, Friis H, Michaelsen KF. Effect of Probiotics on Diarrhea in Children With Severe Acute Malnutrition: A Randomized Controlled Study in Uganda. J Pediatr Gastroenterol Nutr. 2017 Mar;64(3):396-403. doi: 10.1097/MPG.0000000000001515. PMID 28079729
- [Background] Hock BD, Kato M, McKenzie JL, Hart DN. A soluble form of CD83 is released from activated dendritic cells and B lymphocytes, and is detectable in normal human sera. Int Immunol. 2001 Jul;13(7):959-67. doi: 10.1093/intimm/13.7.959. PMID 11431426
- [Background] Hunt KM, Foster JA, Forney LJ, Schutte UM, Beck DL, Abdo Z, Fox LK, Williams JE, McGuire MK, McGuire MA. Characterization of the diversity and temporal stability of bacterial communities in human milk. PLoS One. 2011;6(6):e21313. doi: 10.1371/journal.pone.0021313. Epub 2011 Jun 17. PMID 21695057
- [Background] Islam MM, Peerson JM, Ahmed T, Dewey KG, Brown KH. Effects of varied energy density of complementary foods on breast-milk intakes and total energy consumption by healthy, breastfed Bangladeshi children. Am J Clin Nutr. 2006 Apr;83(4):851-8. doi: 10.1093/ajcn/83.4.851. PMID 16600938
- [Background] Kerac M, Bunn J, Seal A, Thindwa M, Tomkins A, Sadler K, Bahwere P, Collins S. Probiotics and prebiotics for severe acute malnutrition (PRONUT study): a double-blind efficacy randomised controlled trial in Malawi. Lancet. 2009 Jul 11;374(9684):136-44. doi: 10.1016/S0140-6736(09)60884-9. PMID 19595348
- [Background] Handelsman J, Rondon MR, Brady SF, Clardy J, Goodman RM. Molecular biological access to the chemistry of unknown soil microbes: a new frontier for natural products. Chem Biol. 1998 Oct;5(10):R245-9. doi: 10.1016/s1074-5521(98)90108-9. PMID 9818143
- [Background] Kuroishi T, Tanaka Y, Sakai A, Sugawara Y, Komine K, Sugawara S. Human parotid saliva contains soluble toll-like receptor (TLR) 2 and modulates TLR2-mediated interleukin-8 production by monocytic cells. Mol Immunol. 2007 Mar;44(8):1969-76. doi: 10.1016/j.molimm.2006.09.028. Epub 2006 Nov 1. PMID 17081611
- [Background] Lepage P, Leclerc MC, Joossens M, Mondot S, Blottiere HM, Raes J, Ehrlich D, Dore J. A metagenomic insight into our gut's microbiome. Gut. 2013 Jan;62(1):146-58. doi: 10.1136/gutjnl-2011-301805. Epub 2012 Apr 23. PMID 22525886
- [Background] LeBouder E, Rey-Nores JE, Rushmere NK, Grigorov M, Lawn SD, Affolter M, Griffin GE, Ferrara P, Schiffrin EJ, Morgan BP, Labeta MO. Soluble forms of Toll-like receptor (TLR)2 capable of modulating TLR2 signaling are present in human plasma and breast milk. J Immunol. 2003 Dec 15;171(12):6680-9. doi: 10.4049/jimmunol.171.12.6680. PMID 14662871
- [Background] Human Microbiome Project Consortium. A framework for human microbiome research. Nature. 2012 Jun 13;486(7402):215-21. doi: 10.1038/nature11209. PMID 22699610
- [Background] Panigrahi P, Parida S, Nanda NC, Satpathy R, Pradhan L, Chandel DS, Baccaglini L, Mohapatra A, Mohapatra SS, Misra PR, Chaudhry R, Chen HH, Johnson JA, Morris JG, Paneth N, Gewolb IH. A randomized synbiotic trial to prevent sepsis among infants in rural India. Nature. 2017 Aug 24;548(7668):407-412. doi: 10.1038/nature23480. Epub 2017 Aug 16. PMID 28813414
- [Background] Prata MM, Havt A, Bolick DT, Pinkerton R, Lima A, Guerrant RL. Comparisons between myeloperoxidase, lactoferrin, calprotectin and lipocalin-2, as fecal biomarkers of intestinal inflammation in malnourished children. J Transl Sci. 2016;2(2):134-139. doi: 10.15761/JTS.1000130. Epub 2016 Mar 25. PMID 27746954
- [Background] Roudkenar MH, Kuwahara Y, Baba T, Roushandeh AM, Ebishima S, Abe S, Ohkubo Y, Fukumoto M. Oxidative stress induced lipocalin 2 gene expression: addressing its expression under the harmful conditions. J Radiat Res. 2007 Jan;48(1):39-44. doi: 10.1269/jrr.06057. Epub 2007 Jan 16. PMID 17229997
- [Background] Shendure J, Ji H. Next-generation DNA sequencing. Nat Biotechnol. 2008 Oct;26(10):1135-45. doi: 10.1038/nbt1486. PMID 18846087
- [Background] Sheridan PO, Bindels LB, Saulnier DM, Reid G, Nova E, Holmgren K, O'Toole PW, Bunn J, Delzenne N, Scott KP. Can prebiotics and probiotics improve therapeutic outcomes for undernourished individuals? Gut Microbes. 2014 Jan-Feb;5(1):74-82. doi: 10.4161/gmic.27252. Epub 2013 Dec 16. PMID 24637591
- [Background] Smilowitz JT, Moya J, Breck MA, Cook C, Fineberg A, Angkustsiri K, Underwood MA. Safety and tolerability of Bifidobacterium longum subspecies infantis EVC001 supplementation in healthy term breastfed infants: a phase I clinical trial. BMC Pediatr. 2017 May 30;17(1):133. doi: 10.1186/s12887-017-0886-9. PMID 28558732
- [Background] Tringe SG, von Mering C, Kobayashi A, Salamov AA, Chen K, Chang HW, Podar M, Short JM, Mathur EJ, Detter JC, Bork P, Hugenholtz P, Rubin EM. Comparative metagenomics of microbial communities. Science. 2005 Apr 22;308(5721):554-7. doi: 10.1126/science.1107851. PMID 15845853
- [Background] Wang WL, Xu SY, Ren ZG, Tao L, Jiang JW, Zheng SS. Application of metagenomics in the human gut microbiome. World J Gastroenterol. 2015 Jan 21;21(3):803-14. doi: 10.3748/wjg.v21.i3.803. PMID 25624713
- [Background] Williams JE, Price WJ, Shafii B, Yahvah KM, Bode L, McGuire MA, McGuire MK. Relationships Among Microbial Communities, Maternal Cells, Oligosaccharides, and Macronutrients in Human Milk. J Hum Lact. 2017 Aug;33(3):540-551. doi: 10.1177/0890334417709433. Epub 2017 Jun 13. PMID 28609134
- [Background] Woese CR, Fox GE. Phylogenetic structure of the prokaryotic domain: the primary kingdoms. Proc Natl Acad Sci U S A. 1977 Nov;74(11):5088-90. doi: 10.1073/pnas.74.11.5088. PMID 270744
- [Derived] Nuzhat S, Palit P, Mahfuz M, Islam MR, Hasan SMT, Islam MM, Sarker SA, Kyle DJ, Flannery RL, Vinjamuri A, Lebrilla CB, Ahmed T. Association of human milk oligosaccharides and nutritional status of young infants among Bangladeshi mother-infant dyads. Sci Rep. 2022 Jun 8;12(1):9456. doi: 10.1038/s41598-022-13296-w. PMID 35676397